CLINICAL TRIAL: NCT05559255
Title: Changes in Pain, Spasticity, and Quality of Life After Use of Counterstrain Osteopathic Manipulative Treatment in Individuals With Spinal Cord Injury
Brief Title: Changes in Pain, Spasticity, and Quality of Life After Use of Counterstrain Treatment in Individuals With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Carey University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, David Dolbow, David R. Dolbow, Primary Investigator, William Carey University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WilliamCareyU-COM-PT
Record Dates: First submitted 2022-08-10; First posted 2022-09-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pain; Spasticity, Muscle; Quality of Life
Keywords: pain; spasticity; quality of life; spinal cord injury; counterstrain manual manipulative treatment
MeSH Terms: conditions — Pain; Muscle Spasticity; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Thirty individuals with pain and spasticity after SCI will undergo the counterstrain manual manipulative treatment three times per week for four weeks. Pre and post program measures for pain, spasticity, and quality of life will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Counterstrain manual manipulative treatment — The steps required to perform counterstrain in any region of the body are as follows:
  1. Find the tender point.
  2. Assess the tenderness using a pain scale.
  3. Passively and gently place the patient in a position-of-comfort that results in the greatest reduction of tenderness at the tender point. Approximate the position first, then fine-tune through small arcs of movement. Aim to achieve at least 70% tenderness reduction, with the goal of 100%.
  4. Maintain the position for 90 seconds while continuing to monitor the patient's tender point.
  5. Passively return the patient to a neutral position.
  6. Re-test for tenderness at the tender point.

SUMMARY:
Individuals with spinal cord injury (SCI) often suffer from pain and spasticity. Traditional treatments for both of these conditions have been medications. However, it has been suggested that the counterstrain osteopathic manual manipulation treatment can decrease pain and possibly spasticity. The aim of this study is to investigate the effects of counterstrain osteopathic manual manipulation treatment on pain and spasticity in individuals with SCI.

DETAILED DESCRIPTION:
Individuals with SCI often suffer from pain and spasticity. Traditional treatments for both of these conditions have been medications. However, it has been suggested that the counterstrain osteopathic manual manipulation treatment can decrease pain and possibly spasticity. The aim of this study is to investigate the effects of counterstrain osteopathic manual manipulation treatment on pain and spasticity in individuals with SCI.

The hypothesis for our research aim is that the use of the counterstrain osteopathic manipulation treatment will decrease pain, decrease muscle spasticity, and improve the participants' perception of their quality of life. After reviewing and signing an informed consent form that has been approved by the institutional review board at William Carey University, each participant will then provide a signed clearance form from their primary care physician stating that they have been screened and are approved to participate in the study. Participants will be asked to attend the William Carey Research Laboratory for the initial pre-testing. Height, weight, age, level of injury, and time since the injury will be recorded during the first visit to the William Carey University Research Laboratory. Vital signs including heart rate, blood pressure, and oxygen saturation will be assessed before and after the counterstrain technique is performed to ensure hemodynamic stability. The participants will be monitored by a licensed osteopathic medical physician. Any indication of discomfort by the participant will be evaluated which includes tests pertaining to pain, spasticity, and quality of life. Tests including the Universal Pain Assessment Tool (UPAT), Douleur Neuropathique 4 (DN4) Neuropathic Pain Diagnostic Questionnaire, and Spinal Cord Injury Spasticity Evaluation Tool will be performed while the participants are seated in their wheelchairs before and after each session. The Modified Ashworth Test will be performed both while the patient is seated and again while supine on the treatment table prior to and after each session. The World Health Organization Brief Quality of Life Questionnaire will be performed while the participants are seated in their wheelchairs at the start of the four-week program and then again after the four-week program has ended.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with C4-L5 spinal cord injury
* American Spinal Injury Association Impairment Scale A, B, and C as per International Standards for Neurological Classification of spinal cord injury.
* Participants will be one or more years post-injury
* Age 21-70 years

Exclusion Criteria:

* Pressure wounds on buttocks or feet
* Unhealed bone fractures or history of fragility fractures
* Uncontrolled cardiovascular or metabolic disease
* Diagnosed with severe osteoporosis (T score ≤ 4)
* Uncontrolled autonomic dysreflexia.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Neurogenic Pain after each session | Sessions/days 1,2,3,4,5,6,7,8,9,10,11,12
  Pain as described by the participant ( Universal Pain Assessment Tool (UPAT), score range from 0-10 where 0 is no pain and 10 is the worst pain possible.
Muscle Spasticity | Sessions/days 1,2,3,4,5,6,7,8,9,10,11,12
  Spasticity as described by the participants' Modified Ashworth Test scores 0-4 where 0 is no tone and 4 is rigid tone.
Self-perceived quality of life via WHO Brief QoL questionnaire | four weeks (sessions 1 and 12)
  Quality of life as described by the participants (World Health Organization Quality of Life questionnaire) Twenty six questions each with a Likert scale range 1-5 where 1 equals not at all and 5 equals extremely. Five is typically the better score.
Change in neuropathic pain after the 4 weeks of the program. | four weeks (sessions 1 and 12)
  The Neuropathic Pain Diagnostic Questionnaire). Ten yes or no questions without a numerical score. Then six questions concerning the impact of pain on life activities with a 0-10 scale where 0 is "does not interfere" and 10 is "completely interferes"

CONTACTS AND LOCATIONS:
Overall Officials: Italo Subbarao, DO, Study Director — William Carey University
Locations (1):
- William Carey University, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available.